CLINICAL TRIAL: NCT00993109
Title: Randomized,Open-label,Parallel Design Comparator Study of Effect of Nifedipine GITS/OROS (Adalat) 30 mg in Combination With Valsartan (Diovan) 80 mg Compared to Valsartan (Diovan) 160 mg Monotherapy in Patients Whose Blood Pressure is Not Well Controlled by Valsartan 80 mg Alone
Brief Title: Low-dose Nifedipine-Valsartan Combination Compared to Up-titrated Valsartan Monotherapy in Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14511; ADVISE (Other: Company Internal)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
Keywords: Nifedipine GITS/OROS (Adalat®); Valsartan (Diovan®); Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Adalat (Nifedipine, BAYA1040)
- Arm 2 (Active Comparator)
  Interventions: Drug: Diovan (Valsartan)

INTERVENTIONS:
Drug: Adalat (Nifedipine, BAYA1040) — Nifedipine GITS/OROS 30 mg OM + Valsartan 80 mg OM
  Arms: Arm 1
Drug: Diovan (Valsartan) — Valsartan 160 mg OM (Two Valsartan 80mg tablets)
  Arms: Arm 2

SUMMARY:
This will be a multi-center, prospective, randomized, open-label, parallel design, two arm comparator trial. In the proposed study, the investigators will compare low-dose combination therapy of Nifedipine GITS/OROS plus Valsartan with up-titrated monotherapy of Valsartan with respect to their blood pressure-decreasing effects in patients with essential hypertension.The study consists of a screening visit, followed by randomization and administration of either Nifedipine GITS/OROS 30 mg in combination with Valsartan 80 mg or Valsartan 160 mg for 12 weeks of treatment.The primary efficacy parameters will be mean SBP and DBP on office BP monitoring at 12 weeks of treatment compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 75 years
* Essential hypertension not well controlled by current low dose (80 mg) valsartan monotherapy for at least 4 weeks. Patients on prior treatment with monotherapy diuretic, ACE-I or beta blocker or an ARB other than valsartan and switched to the current low dose valsartan 80 mg monotherapy for at least 4 weeks are also eligible, provided the hypertension is still not well controlled.
* Office systolic blood pressure (sitting) >140 mmHg (sitting for >/= 5 min., no cigarettes and/or coffee/tea for >/=30 min. before BP measurement).
* BMI <33 kg/m2

Exclusion Criteria:

* Participation in any clinical investigational drug study within the previous 12 weeks
* Concomitant treatments with:

  1. Any anti-hypertensive treatment other than Valsartan 80 mg
  2. Cytochrome P450-3A4 inhibitors or inducers
  3. Potassium-sparing diuretics
* Severe hypertension (DBP >/= 110 mm Hg and/or SBP >/= 180 mm Hg) and/or evidence of secondary forms of hypertension
* Any of the following cardiovascular diseases:
* History of cardiovascular shock
* Myocardial infarction or unstable angina within the previous 6 months
* Severe cardiac valve disease
* Past or present severe rhythm or conduction disorder.
* Cerebrovascular ischemic event and/or history of intracerebral hemorrhage or subarachnoid hemorrhage (SAH) within the previous 12 months
* Type 1 or 2 diabetes mellitus
* Proteinuria
* Uncorrected hypokalemia or hyperkalemia, sodium depletion and/or hypovolemia
* Gastrointestinal disease resulting in the potential for malabsorption and/or severe gastro-intestinal tract narrowing; kock pouch (ileostomy after proctocolectomy)
* Cholestasis or biliary obstruction
* Liver disease or aspartate aminotransferase (AST) / alanine aminotransferase (ALT) levels >3 x upper limits of normal (ULN)
* Renal failure, creatinine level >2.0 mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean Systolic BP and Diastolic BP on office Blood Pressure monitoring | Baseline and 12 weeks of treatment

SECONDARY OUTCOMES:
Response rate (>/=10mmHg decrease of office SBP and >/=5mmHg decrease of office DBP) | 8 and 12 weeks of treatment
Control rate (</=140/90 of office BP) | 8 and 12 weeks of treatment
Change in pulse pressure (difference between SBP and DBP) | 12 weeks of treatment
Reduction in Urinary microalbumin excretion(UAE) in patients with microalbuminuria | Baseline and 12 weeks of treatment
Adverse Event reporting | At the start, every 4 weeks during treatment and at the end of treatment
Vitals signs | At the start, every 4 weeks during treatment and at the end of treatment
Laboratory tests | At the start and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- China (7):
  - Guangzhou, Guangdong
  - Shijiazhuang, Hebei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Shenyang, Liaoning
  - Beijing
  - Shanghai
- South Korea (6):
  - Donggu, Gwangju Gwang''yeogsi
  - Bucheon-si, Gyeonggido
  - Yangsan, Gyeongsangnam-do
  - Jongno-gu
  - Junggu
  - Seoul

REFERENCES:
- [Derived] Ke YN, Dong YG, Ma SP, Yuan H, Ihm SH, Baek SH; ADVISE study group. Improved blood pressure control with nifedipine GITS/valsartan combination versus high-dose valsartan monotherapy in mild-to-moderate hypertensive patients from Asia: results from the ADVISE study, a randomized trial. Cardiovasc Ther. 2012 Dec;30(6):326-32. doi: 10.1111/1755-5922.12003. PMID 23134522